CLINICAL TRIAL: NCT01295697
Title: A Phase 1/2 Study of EZN-2208 in Children, Adolescents, and Young Adults With Relapsed or Refractory Solid Tumors
Brief Title: Study of EZN-2208 Pediatric Patients With Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Program suspended and divested
Sponsor: Enzon Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EZN-2208-05
Record Dates: First submitted 2010-12-03; First posted 2011-02-14 (Estimated); Last update posted 2022-02-14 (Actual); Status verified 2012-03

CONDITIONS: Solid Tumors
Keywords: Patients with non-CNS or CNS tumors; Pediatric patients with Relapsed/Refractory Solid Tumors
MeSH Terms: conditions — Central Nervous System Neoplasms | interventions — EZN-2208

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EZN-2208 (Experimental): Cytotoxic Agent
  Interventions: Drug: EZN-2208

INTERVENTIONS:
Drug: EZN-2208 — Experimental
  Other Names: PEG-SN38

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of EZN-2208 that can be given to pediatric patients with Relapsed or Refractory Solid Tumors. The safety of the study drug and its effect on the disease will also be studied.

DETAILED DESCRIPTION:
Pharmacokinetic (PK) testing of EZN-2208, will be performed for patients who volunteer. PK testing measures the amount of a drug in the body at different time points.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologic verification of malignancy at original diagnosis or relapse.
* Measurable or evaluable disease
* Karnofsky score more or equal to 50 for patients >16 years of age and Lansky score more or equal to 50 for patients <16 years of age
* Patients previously treated with irinotecan will be eligible for this study if they have not had documented progressive disease during treatment with an irinotecan-containing regimen.
* Adequate hematologic, hepatic, coagulation, renal, and metabolic function

Exclusion Criteria:

* Pregnant or breast feeding patients will not be enrolled in this study
* Patients who are currently receiving other anticancer agents
* Patients who have an uncontrolled infection
* Patients requiring cytochrome P450 3A4 enzyme inducing or inhibiting agents

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2010-02; Primary Completion 2012-08 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Determine the MTD and recommended phase 2 dose of i.v. EZN-2208 administered q3wk. | 2 years
  The study will measure incidence, severity and duration of adverse events graded by NCI CTCAE during first cycle of therapy to determine the MTD.
  A Phase 2 Dose will be recommended by study investigators after considering the frequency and severity of adverse events and the ability to maintain dose schedule

SECONDARY OUTCOMES:
Assess evidence of tumor response activity of EZN-2208 | 2 years
  An evaluation of objective Tumor response by radiographic scans will be performed every two cycles following the criteria of RECIST 1.1.
Evaluate the safety and tolerability of EZN-2208 | 2 years
  The incidence, severity and duration of adverse events graded by NCI CTCAE during all cycles of therapy will be used to assess safety and tolerability.
Assess the PK profile of EZN-2208 | 2 years
  The pharmacokinetics of EZN-2208 will be established by measuring the concentration of EZN-2208 and SN-38 over time in patient blood samples.

CONTACTS AND LOCATIONS:
Overall Officials: Rochelle Bagatell, MD, Study Chair — Developmental Therapeutics Program, The Children's Hospital of Philadelphia, CTRB 4022; 3501 Civic Center Blvd. Philadelphia, PA 19104
Locations (4):
- United States (4):
  - Lia Gore, MD, Aurora, Colorado
  - Suzanne Shusterman, MD, Boston, Massachusetts
  - Rochelle Bagatell, MD (Principal Investigator), Philadelphia, Pennsylvania
  - Jodi Muscal, MD, Houston, Texas